CLINICAL TRIAL: NCT00205556
Title: Effect of Increased Convective Clearance by On-line Hemodiafiltration on All Cause and Cardiovascular Mortality in Chronic Hemodialysis Patients: The Dutch Convective Transport Study (CONTRAST)
Brief Title: Effect of Increased Convective Clearance by On-Line Hemodiafiltration on All Cause Mortality in Chronic Hemodialysis Patients
Acronym: CONTRAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: UMC Utrecht (Other); Medical Center Alkmaar (Other); Maasstad Hospital (Other); Julius Center for Health Sciences and Primary Care, Utrecht (Unknown); Dutch Kidney Foundation (Other); Fresenius Medical Care North America (Industry); Gambro Renal Products, Inc. (Industry); Baxter Healthcare Corporation (Industry); Roche Pharma AG (Industry)
Responsible Party: contact person: MPC Grooteman MD PhD, Vrije Universiteit Medical Center and University Medical Center Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METC VUmc 03/097; ISRCTN38365125; CCMO number P03.1089L; Dutch Kidney Found C 02.2019
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: End-stage Renal Disease; Cardiovascular Disease
Keywords: online hemodiafiltration; low flux hemodialysis; cardiovascular disease; endothelial dysfunction; uremic toxicity; quality of life; nutritional status
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: low flux hemodialysis (Other): standard treatment
  Interventions: Procedure: low flux hemodialysis
- 2 on-line hemodiafiltration (Active Comparator)
  Interventions: Procedure: on-line hemodiafiltration

INTERVENTIONS:
Procedure: on-line hemodiafiltration — addition of convective transport to regular dialysis treatment by using on-line hemodiafiltration
  Arms: 2 on-line hemodiafiltration
Procedure: low flux hemodialysis — standard treatment
  Arms: 1: low flux hemodialysis

SUMMARY:
The purpose of this study is to compare the effect of low flux hemodialysis with online hemodiafiltration on all cause mortality and a combination of cardiovascular morbidity and mortality in chronic hemodialysis patients.

DETAILED DESCRIPTION:
Today, an increasing number of patients with chronic renal failure (CRF) is treated with (on-line) hemodiafiltration (HDF). This practice is based on the assumption that the high incidence of cardiovascular (CV) disease, as observed in patients with CRF, is at least partially related to the retention of uremic toxins in the middle and large-middle molecular (MM) range. As HDF lowers these molecules more effectively than HD, it has been suggested that this treatment improves CV outcome, if compared to standard HD.

Thus far, no definite data on the effects of HDF on CV parameters and/or clinical end-points are available. Promising data include a reduction of left ventricular mass index (LVMi) after one year of treatment with acetate free bio-filtration (AFB). Furthermore, relatively high survival rates were reported in a single center non-experimental study on patients who were treated with HDF, if compared to the EDTA registry data on HD-treated patients. Yet, these data are of observational nature, with the possibility of being biased by confounding by indication.

As the accumulation of MMW substances has been implicated in increased oxidative stress and endothelial dysfunction, a reduction of these compounds might improve these derangements. In addition, cardiac dysfunction, atherosclerosis (as measured by left ventricular mass index [LVMi], carotid intima media thickness [CIMT]) and vascular stiffness (as measured by pulse wave velocity [PWV]) might be reduced during HDF, as compared to low-flux HD.

Therefore, we propose a prospective, randomized multicenter trial, comparing (on-line) HDF with HD. After a stabilization period, an expected number of 700 chronic HD patients will be randomized to either HDF or low-flux HD and followed during 1-6 years. Primary end points are all cause mortality and combined CV events and mortality. In addition, LVMi, PWV, CIMT and various parameters of oxidative stress, acute phase reaction (APR) and endothelial function will be assessed and compared between treatment groups.

This study will provide strong evidence on the efficacy of HDF compared to low flux HD on CV morbidity and mortality, which is currently lacking but urgently needed. It is highly likely that the outcome of this study will affect current clinical practice considerably, in the Netherlands as well as internationally. Moreover, the study will point towards the mechanisms underlying the effects of HDF.

The following hypotheses will be tested:

1. All-cause mortality and combined CV morbidity and mortality in patients treated with (on-line) HDF is lower than in patients treated with standard low-flux HD.
2. A reduction in MMW uremic toxins by HDF leads to an improvement of the 'uremic profile' (as measured by AGE-levels, homocysteine levels, oxidative stress, and endothelial dysfunction), if compared to standard low-flux HD.
3. The improvement of the 'uremic profile' in HDF-treated patients results in an improvement of endothelial function with a reduction in the progression of vascular injury (as measured by CIMT and PWV) and a reduction in LVMi, if compared to standard low-flux HD.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by HD 2 or 3 times a week, for at least 2 months
* Patients able to understand the study procedures
* Patients willing to provide written informed consent

Exclusion Criteria:

* Current age < 18 years
* Treatment by HDF or high flux HD in the preceding 6 months
* Severe incompliance (severe non-adherence to the dialysis procedure and accompanying prescriptions, especially frequency and duration of dialysis treatment and fluid restriction)
* Life expectancy < 3 months due to non renal disease
* Participation in other clinical intervention trials evaluating cardiovascular outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2004-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
all cause mortality | entire follow up (until dead or end of study, 1-7 years)

SECONDARY OUTCOMES:
fatal and non-fatal cardiovascular events | entire follow up (until death or end of study, 1-7 years)
Left ventricular mass index (LVMi), carotid IMT (intima media thickness), aortic pulse wave velocity (PWV) | first 3 years
laboratory markers of endothelial dysfunction, micro-inflammation, oxidative stress | first three years of follow up
lipid profiles, uremic toxins | first three years
quality of life | entire follow up (until death or end of study, 1-7 years)
nutritional state | entire follow up (until death or end of study 1-7 years)
anemia management | first 12 months of follow up
  hemoglobin levels, erythropoietin use / resistance iron saturation / ferritin levels, prescription of iron medication
cost utility analysis | entire follow up (until death or end of study, 1-7 years)
hospital admissions | entire follow up (until death or end of study, 1-7 years)
  hospitalization days hospital admission for infections hospital admission for any cause
blood pressure and antihypertensive medication | entire follow up (until death or end of study, 1-7 years)
residual kidney function | entire follow up (until death or end of study, 1-7 years)
mineral bone disease | entire follow up (until death or end of study, 1-7 years)
  laboratory parameters of mineral bone disease and medication (phosphate binders, vitamin D (or analogues), cinacalet)
parameters of treatment / treatment delivery | entire follow up (until death or end of study, 1-7 years)
  dialysis efficiency (Kt/V urea); bloodflow, dialysate flow, ultrafiltration volume, (HDF:) convection volume

CONTACTS AND LOCATIONS:
Overall Officials: Menso J Nubé, MD PhD, Study Director — Medical Center Alkmaar; Piet M ter Wee, MD PhD, Study Chair — Vrije Universiteit Medical Center, Amsterdam; Peter J Blankestijn, MD PhD, Study Chair — Universityr Medical Center Utrecht; René A van den Dorpel, MD PhD, Study Director — Medisch Centrum Rijnmond Zuid - locatie Clara, Rotterdam; Michiel L Bots, MD PhD, Study Director — Julius Center for Health Sciences and Primary Care, Utrecht; Muriel PC Grooteman, MD PhD, Principal Investigator — Vrije Universiteit Medical Center, Amsterdam
Locations (29):
- Canada (2):
  - Dr Georges-L. Dumont Regional Hospital, Moncton, New Brunswick
  - Centre Hospitalier de L'Université de Montreal, Hopital Notre Dame, Montreal
- Netherlands (26):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Medisch Centrum Alkmaar, Alkmaar
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academical Medical Center, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Dialyse Kliniek Noord, Beilen
  - Slingeland Ziekenhuis, Doetinchem
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Oosterscheldeziekenhuis, Goes
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Rijnland Ziekenhuis, Leiderdorp
  - University Medical Center St Radboud, Nijmegen
  - Franciscus Ziekenhuis, Roosendaal
  - Sint Franciscus Gasthuis, Rotterdam
  - Medisch Centrum Rijnmond Zuid - locatie Clara, Rotterdam
  - Orbis Medisch en Zorgcentrum, Sittard
  - Ziekenhuis Zeeuws-Vlaanderen, Terneuzen
  - Haga Ziekenhuis (locatie Leyenburg), The Hague
  - St Elisabeth Ziekenhuis, Tilburg
  - Stichting Dianet, Utrecht
  - University Medical Center Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - Isala Klinieken, Zwolle
- Haukeland Universitetssykehus, Bergen, Norway

REFERENCES:
- [Background] Penne EL, Blankestijn PJ, Bots ML, van den Dorpel MA, Grooteman MP, Nube MJ, van der Tweel I, Ter Wee PM; the CONTRAST study group. Effect of increased convective clearance by on-line hemodiafiltration on all cause and cardiovascular mortality in chronic hemodialysis patients - the Dutch CONvective TRAnsport STudy (CONTRAST): rationale and design of a randomised controlled trial [ISRCTN38365125]. Curr Control Trials Cardiovasc Med. 2005 May 20;6(1):8. doi: 10.1186/1468-6708-6-8. PMID 15907201
- [Background] Penne EL, Blankestijn PJ, Bots ML, van den Dorpel MA, Grooteman MP, Nube MJ, ter Wee PM; CONTRAST Group. Resolving controversies regarding hemodiafiltration versus hemodialysis: the Dutch Convective Transport Study. Semin Dial. 2005 Jan-Feb;18(1):47-51. doi: 10.1111/j.1525-139X.2005.18107.x. PMID 15663765
- [Background] Penne EL, Blankestijn PJ, Bots ML, van den Dorpel MA, Grooteman MP, Nube MJ, ter Wee PM. [New study evaluating online haemodiafiltration for the reduction of cardiovascular morbidity and mortality in patients undergoing chronic haemodialysis]. Ned Tijdschr Geneeskd. 2006 Jul 15;150(28):1583-5. Dutch. PMID 16886698
- [Background] van der Weerd NC, Penne EL, van den Dorpel MA, Grooteman MP, Nube MJ, Bots ML, ter Wee PM, Blankestijn PJ. Haemodiafiltration: promise for the future? Nephrol Dial Transplant. 2008 Feb;23(2):438-43. doi: 10.1093/ndt/gfm791. Epub 2007 Nov 28. No abstract available. PMID 18045819
- [Background] Penne EL, van Berkel T, van der Weerd NC, Grooteman MP, Blankestijn PJ. Optimizing haemodiafiltration: tools, strategy and remaining questions. Nephrol Dial Transplant. 2009 Dec;24(12):3579-81. doi: 10.1093/ndt/gfp333. Epub 2009 Jul 13. No abstract available. PMID 19596741
- [Background] van der Weerd NC, Penne EL, Grooteman MP. Effect of hemofiltration on mortality: no definite answer yet. Am J Kidney Dis. 2009 Mar;53(3):562-3; author reply 563. doi: 10.1053/j.ajkd.2008.09.029. No abstract available. PMID 19231743
- [Background] Penne EL, Visser L, van den Dorpel MA, van der Weerd NC, Mazairac AH, van Jaarsveld BC, Koopman MG, Vos P, Feith GW, Kremer Hovinga TK, van Hamersvelt HW, Wauters IM, Bots ML, Nube MJ, Ter Wee PM, Blankestijn PJ, Grooteman MP. Microbiological quality and quality control of purified water and ultrapure dialysis fluids for online hemodiafiltration in routine clinical practice. Kidney Int. 2009 Sep;76(6):665-72. doi: 10.1038/ki.2009.245. Epub 2009 Jul 15. PMID 19606080
- [Background] den Hoedt CH, Mazairac AHA, van den Dorpel MA, Grooteman MPC, Blankestijn PJ. Effect of hemodiafiltration on mortality, inflammation and quality of life. Contrib Nephrol. 2011;168:39-52. doi: 10.1159/000321743. Epub 2010 Oct 7. PMID 20938124
- [Result] Penne EL, van der Weerd NC, Bots ML, van den Dorpel MA, Grooteman MP, Levesque R, Nube MJ, Ter Wee PM, Blankestijn PJ; CONTRAST investigators. Patient- and treatment-related determinants of convective volume in post-dilution haemodiafiltration in clinical practice. Nephrol Dial Transplant. 2009 Nov;24(11):3493-9. doi: 10.1093/ndt/gfp265. Epub 2009 Jun 10. PMID 19515802
- [Result] Penne EL, van der Weerd NC, van den Dorpel MA, Grooteman MP, Levesque R, Nube MJ, Bots ML, Blankestijn PJ, ter Wee PM; CONTRAST Investigators. Short-term effects of online hemodiafiltration on phosphate control: a result from the randomized controlled Convective Transport Study (CONTRAST). Am J Kidney Dis. 2010 Jan;55(1):77-87. doi: 10.1053/j.ajkd.2009.09.023. Epub 2009 Dec 5. PMID 19962805
- [Result] Mazairac AH, de Wit GA, Penne EL, van der Weerd NC, Grooteman MP, van den Dorpel MA, Nube MJ, Buskens E, Levesque R, Ter Wee PM, Bots ML, Blankestijn PJ; CONTRAST investigators. Protein-energy nutritional status and kidney disease-specific quality of life in hemodialysis patients. J Ren Nutr. 2011 Sep;21(5):376-386.e1. doi: 10.1053/j.jrn.2010.08.004. Epub 2010 Dec 30. PMID 21194971
- [Result] Penne EL, van der Weerd NC, Grooteman MP, Mazairac AH, van den Dorpel MA, Nube MJ, Bots ML, Levesque R, ter Wee PM, Blankestijn PJ; CONTRAST investigators. Role of residual renal function in phosphate control and anemia management in chronic hemodialysis patients. Clin J Am Soc Nephrol. 2011 Feb;6(2):281-9. doi: 10.2215/CJN.04480510. Epub 2010 Oct 28. PMID 21030579
- [Result] Penne EL, van der Weerd NC, Blankestijn PJ, van den Dorpel MA, Grooteman MP, Nube MJ, Ter Wee PM, Levesque R, Bots ML; CONTRAST investigators. Role of residual kidney function and convective volume on change in beta2-microglobulin levels in hemodiafiltration patients. Clin J Am Soc Nephrol. 2010 Jan;5(1):80-6. doi: 10.2215/CJN.03340509. Epub 2009 Nov 12. PMID 19965537
- [Result] Mazairac AH, de Wit GA, Grooteman MP, Penne EL, van der Weerd NC, van den Dorpel MA, Nube MJ, Levesque R, Ter Wee PM, Bots ML, Blankestijn PJ; CONTRAST investigators. A composite score of protein-energy nutritional status predicts mortality in haemodialysis patients no better than its individual components. Nephrol Dial Transplant. 2011 Jun;26(6):1962-7. doi: 10.1093/ndt/gfq643. Epub 2010 Oct 14. PMID 20947533
- [Result] Mazairac AH, de Wit GA, Penne EL, van der Weerd NC, de Jong B, Grooteman MP, van den Dorpel MA, Buskens E, Dekker FW, Nube MJ, Ter Wee PM, Boeschoten EW, Bots ML, Blankestijn PJ; CONTRAST investigators. Changes in quality of life over time--Dutch haemodialysis patients and general population compared. Nephrol Dial Transplant. 2011 Jun;26(6):1984-9. doi: 10.1093/ndt/gfq680. Epub 2010 Nov 4. PMID 21051503
- [Derived] de Roij van Zuijdewijn CL, Ter Wee PM. Assessment of Protein-Energy Wasting: Quest for the Gold Standard. J Ren Nutr. 2016 May;26(3):204-5. doi: 10.1053/j.jrn.2016.01.012. Epub 2016 Feb 20. No abstract available. PMID 26908190
- [Derived] de Roij van Zuijdewijn CL, Grooteman MP, Bots ML, Blankestijn PJ, Steppan S, Buchel J, Groenwold RH, Brandenburg V, van den Dorpel MA, Ter Wee PM, Nube MJ, Vervloet MG. Serum Magnesium and Sudden Death in European Hemodialysis Patients. PLoS One. 2015 Nov 23;10(11):e0143104. doi: 10.1371/journal.pone.0143104. eCollection 2015. PMID 26600017
- [Derived] de Roij van Zuijdewijn CL, Grooteman MP, Bots ML, Blankestijn PJ, van den Dorpel MA, Nube MJ, ter Wee PM. Comparing Tests Assessing Protein-Energy Wasting: Relation With Quality of Life. J Ren Nutr. 2016 Mar;26(2):111-7. doi: 10.1053/j.jrn.2015.09.003. Epub 2015 Oct 23. PMID 26584787
- [Derived] den Hoedt CH, Grooteman MP, Bots ML, Blankestijn PJ, van der Tweel I, van der Weerd NC, Penne EL, Mazairac AH, Levesque R, ter Wee PM, Nube MJ, van den Dorpel MA; CONTRAST investigators. The Effect of Online Hemodiafiltration on Infections: Results from the CONvective TRAnsport STudy. PLoS One. 2015 Aug 19;10(8):e0135908. doi: 10.1371/journal.pone.0135908. eCollection 2015. PMID 26288091
- [Derived] van der Weerd NC, Den Hoedt CH, Blankestijn PJ, Bots ML, van den Dorpel MA, Levesque R, Mazairac AH, Nube MJ, Penne EL, ter Wee PM, Grooteman MP; CONTRAST Investigators. Resistance to erythropoiesis stimulating agents in patients treated with online hemodiafiltration and ultrapure low-flux hemodialysis: results from a randomized controlled trial (CONTRAST). PLoS One. 2014 Apr 17;9(4):e94434. doi: 10.1371/journal.pone.0094434. eCollection 2014. PMID 24743493
- [Derived] van der Weerd NC, Grooteman MP, Blankestijn PJ, Mazairac AH, van den Dorpel MA, den Hoedt CH, Nube MJ, Penne EL, van der Tweel I, Ter Wee PM, Bots ML; CONTRAST investigators. Poor compliance with guidelines on anemia treatment in a cohort of chronic hemodialysis patients. Blood Purif. 2012;34(1):19-27. doi: 10.1159/000338919. Epub 2012 Aug 8. PMID 22889943